CLINICAL TRIAL: NCT03916380
Title: Assessment of the Intestinal CYP3A Contribution to Drug Interactions With Envarsus XR Using Grapefruit Juice
Brief Title: Drug Interaction With Envarsus XR and Grapefruit Juice
Status: Completed | Type: Observational
Sponsor: Shirley M. Tsunoda (Other)
Responsible Party: Sponsor-Investigator, Shirley M. Tsunoda, Prinicipal Investigator, University of California, San Diego
Organization: University of California, San Diego (Other)
Other Study IDs: 190617
Record Dates: First submitted 2019-04-10; First posted 2019-04-16 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Kidney Transplant; Complications; Drug Interaction Food
Keywords: Tacrolimus; Grapefruit Juice; CYP3A4; Midazolam; Kidney Transplant

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group A: Tacrolimus Extended Release + Midazolam
  Interventions: Dietary Supplement: Grapefruit Juice
- Group B: Tacrolimus Extended Release + Midazolam + Grapefruit Juice
  Interventions: Dietary Supplement: Grapefruit Juice

INTERVENTIONS:
Dietary Supplement: Grapefruit Juice — Single 8 ounce administration of oral grapefruit juice

SUMMARY:
Transplant patients must take lifelong immunosuppression in order to prevent rejection of their organ. Tacrolimus is the most widely used immnosuppressive agent. Part of the routine education given to patients regarding tacrolimus is that they must avoid many drugs and substances that can interact with tacrolimus so that they don't experience side effects or lack of effect. Patients are told they must avoid readily available substances such as grapefruit juice and St. John's wort. A new once daily formulation of tacrolimus, Envarsus XR, may bypass the place in the gut in which many of these drug interactions occur. We will give kidney transplant patients Envarsus with and without grapefruit juice and measure the effect on blood levels throughout the day. Results from this study will also give us information about the likelihood of other drugs interacting with Envarsus XR.

ELIGIBILITY:
Inclusion Criteria:

* Primary Kidney Transplant Age > 18 years At least 3 months post-transplantation Taking a stable dose of tacrolimus extended release with a target trough of 8-10 ng/mL BMI between 18-32

Exclusion Criteria:

* Multi-organ transplant Concomitant use of mTOR inhibitor Concomitant use of belatacept Concomitant use of medication affecting CYP3A or P-gp History of rejection Hypersensitivity to midazolam Hypersensitivity to Envarsus Active diarrhea or constipation BMI < 18 or > 32

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (18 years and older) recipients of a primary kidney transplant who are at least 3 months post-transplantation. Patients will be enrolled as outpatients in the abdominal transplant clinic. For the pharmacokinetic study days at Visit A and Visit B, patients will be outpatients at the UCSD Clinical and Translational Research Institute (CTRI).
  It is anticipated that we will need to screen approximately 60 patients in order to enroll 20. Since we perform approximately 80-100 kidney transplants per year at UCSD Health, we anticipate enrollment will take 6-10 months. Reasons for patients not participating in the study include: not meeting the inclusion/exclusion criteria; not able or willing to participate in the study because of the time commitment; dropping out. If patients drop out of the study, we will replace them with consecutive patients as they become eligible.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Tacrolimus AUC before and after Grapefruit Juice | 2-4 weeks

SECONDARY OUTCOMES:
Tacrolimus AUC compared to Midazolam AUC | 2-4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- UC San Diego Health, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No